CLINICAL TRIAL: NCT01250821
Title: Gonadotrophin Dosage Using a Threshold Nomogram for Ovulation Induction in WHO Group II Anovulatory Infertility
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Holbaek Sygehus (Other)
Responsible Party: Principal Investigator, Mette Petri Lauritsen, MD, PhD student, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-021459-16
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Anovulation; Infertility
Keywords: Infertility; Anovulation; Ovulation induction
MeSH Terms: conditions — Anovulation; Infertility | interventions — Menotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ovulation induction (Experimental)
  Interventions: Drug: Menopur

INTERVENTIONS:
Drug: Menopur — The medication used in this study is the follicle-stimulating hormone "highly purified human menopausal gonadotrophin" (HP-HMG), Menopur, (Ferring a/s).
  Stimulation with HP-hMG (Menopur) is started on day 2-5 of menstrual bleeding.The HP-hMG starting dose is calculated based on the nomogram predicting the threshold dose. The dose-range is from 75 IU/day to 187.5 IU/day.

SUMMARY:
Ovulation disorders are a common cause of infertility in women. Most of these women can be classified as World Health Organization (WHO) Group II anovulatory patients as they have irregular or absent menstrual cycles but normal serum concentrations of follicle stimulation hormone (FSH) and estradiol.

The purpose of this study is to optimize the low-dose-step-up protocol traditionally used for ovulation induction with follicle-stimulating hormone (FSH) in women with anovulatory infertility WHO Group II.

Previous studies have established that menstrual cycle history, mean ovarian volume and BMI are significant predictors of FSH threshold dose in women with anovulatory infertility WHO Group II undergoing ovulation induction (Nyboe Andersen et al., 2008). A FSH dosage nomogram has been constructed based on these variables.

The aim of this study is to evaluate the clinical use of the nomogram in order to test the use of the variables to determine whether an individualized starting dose of FSH can be used for ovulation induction in anovulatory patients.

It is the hypothesis that an individualized starting dose of gonadotrophin will minimize the disadvantages of the treatment and that the stimulation period of the individualized nomogram-based treatment will be 25% shorter than observed in the standard protocol.

The primary endpoint is the proportion of patients who reach the criteria for hCG-administration within 14 days of Menopur stimulation. The results of the study will be compared with the data obtained in the Menopur Ovulation Induction Trial (Platteau et al., 2006).

ELIGIBILITY:
Inclusion Criteria:

1. Anovulatory infertility
2. Age 18 - 39 years
3. Anovulation with oligomenorrhoea (> 35 days of mean cycle length) or amenorrhoea
4. Normal serum FSH (< 10 IU/l)
5. Two ovaries
6. BMI < 35
7. First FSH/HMG cycle at the Fertility clinic.
8. A sperm sample compatible with conception or semen from a donor.
9. Tubal patency documented by either hysterosalpingography (HSG) or hysterosalpingography by ultrasound (HSU) in cases where the woman has had a pelvic infection or pelvic surgery.

Exclusion Criteria:

1. A history of >12 ovulation induction cycles without achieving pregnancy.
2. More than three earlier gonadotropin cycles at other clinics or earlier treatments with threshold doses below 75.
3. Known hyperprolactinaemia or any other endocrine disturbance or systemic disease of the pituitary gland, thyroid gland, adrenal gland, pancreas, liver or kidney.
4. Undiagnosed vaginal bleeding.
5. Acute or chronic infection with HIV or hepatitis.
6. Persistent ovarian cysts or endometriomas detected by ultrasound.
7. Tumors of the hypothalamus, pituitary gland, breast, adrenal gland or ovary.
8. Pregnancy or lactation.
9. Current or past alcohol or drug abuse.
10. A history of chemo- or radiotherapy.
11. Malformations of reproductive organs incompatible with pregnancy.
12. Hypersensitivity to any trial medication.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who reach the criteria for hCG-administration within 14 days of FSH stimulation. | 14 days of FSH stimulation
  The HCG-criteria is defined as:
  1. One follicle with a diameter of >17 mm or two or three follicles > 15 mm (verified by transvaginal ultrasound).
  2. HCG should not be given if there is no response after 35 days or > 4 follicles > 15 mm (unless converted to IVF/ICSI).
  3. If a patient is seen with one to three follicles of 15 - 16 mms HCG can be administered on the same or on the next day due to a presumed growth of follicles of + 2 mm/day.

SECONDARY OUTCOMES:
Endocrinological characteristics and follicular dynamics of anovulatory infertility WHO Group II | 35 days
  Prediction of FSH response in anovulatory infertility WHO Group II based on endocrinology, sonography, FSH-receptor status and demography

CONTACTS AND LOCATIONS:
Overall Officials: Mette P Lauritsen, MD, Principal Investigator — Rigshospitalet, Denmark; Anders N Andersen, Prof. MD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- The Fertility Clinic, Section 4071, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Nyboe Andersen A, Balen A, Platteau P, Devroey P, Helmgaard L, Arce JC; Bravelle Ovulation Induction (BOI) Study Group. Predicting the FSH threshold dose in women with WHO Group II anovulatory infertility failing to ovulate or conceive on clomiphene citrate. Hum Reprod. 2008 Jun;23(6):1424-30. doi: 10.1093/humrep/den089. Epub 2008 Mar 26. PMID 18372254
- [Background] Platteau P, Andersen AN, Balen A, Devroey P, Sorensen P, Helmgaard L, Arce JC; Menopur Ovulation Induction (MOI) Study Group. Similar ovulation rates, but different follicular development with highly purified menotrophin compared with recombinant FSH in WHO Group II anovulatory infertility: a randomized controlled study. Hum Reprod. 2006 Jul;21(7):1798-804. doi: 10.1093/humrep/del085. Epub 2006 Mar 29. PMID 16571641